CLINICAL TRIAL: NCT06532123
Title: Mechanisms of Improving Fecal Continence Muscles Motor Function in Health and Disease
Brief Title: Mechanisms of Improving Fecal Continence Muscles Motor Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Ling Mei MD, MPH, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO00052310
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: to characterize fatigue characteristic of various continence muscles and to determine the relative/individual contribution of striated continence muscles, including Puborectalis muscle (PRM) and External anal sphincter (EAS) motor function enhancement in improving fecal incontinence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- fatigability of various striated continence muscles healthy adults (Active Comparator): Device: anorectal manometry/vaginal manometry (female) with and without applying c-RED Participants will do repetitive anal contraction and sustained contraction without device and with device in a random order. For contraction with the device, three different resistance level will be applied as described previously.
  For isometric contraction, the annal balloon of the device will be inflated to internal pressure of 500mmHg, which is noncompressible. Participants will repeat the repetitive contraction and sustained contraction.
  Interventions: Device: continence muscles resistance device
- contribution of continence muscles motor function enhancement in improving fecal incontinence (Active Comparator): Device: anorectal manometry/vaginal manometry (female) with c-RED Patients will then be assigned to one of the exercise protocols for 6 weeks. Protocol 1: 20 Kegel like repetitive short contractions against a progressively increased intra-vaginal resistance Protocol 2: 40 Kegel like repetitive short contractions against a progressively increased intra-vaginal resistance Protocol 3: 20 Kegel like repetitive short contractions against a progressively increased intra-anal resistance Protocol 4: 40 Kegel like repetitive short contractions against a progressively increased intra-anal resistance Protocol 5: 20 Kegel like repetitive short contractions without device Protocol 6: 40 Kegel like repetitive short contractions without device Protocol 7: 20 Kegel like repetitive short contractions against the non-compressible balloon as previously mentioned Protocol 8:40 Kegel like repetitive short contractions against the non-compressible balloon as previously mentioned
  Interventions: Device: continence muscles resistance device

INTERVENTIONS:
Device: continence muscles resistance device — The c-RED consists of a noncompliant cylindrical balloon (intra-anal balloon) that is connected to a small compliant balloon (external balloon) by a 2 mm diameter tube and a stopcock to allow for air to be filled and sealed in the system. The system is prefilled with air to determine the amount of air needed for a given internal pressure, or desired resistance of the intra-anal balloon. This is determined using a sphygmomanometer gauge in a sealed system.

SUMMARY:
The investigators hypothesize that different continence muscles have different fatigue characteristics and fatigue induced by resisted contractions will result in significant increase in contractility of the continence muscles and improvement of fecal incontinence severity.

DETAILED DESCRIPTION:
To achieve the specific aim, the investigators will use state-of the-art available techniques and recording modalities, as well as a novel device that provides pre-determined different levels of resistance against contraction of continence muscles to induce measurable fatigue. The investigators will determine and characterize the fatigue characteristics of the striated continence muscles across adult age spectrum and sex. The investigators will determine and compare the effect of 6-weeks daily fatigue on continence musculature motor function and its effect on incontinence severity and related patient quality of life.

Aim1A: the investigators will determine and characterize the fatigue characteristics of the continence muscles induced by repetitive isotonic contractions using various loads, intervals, and repetitions in a. Continence muscle complex (comprised of external anal sphincter muscle group and puborectalis muscle) , and b. puborectalis muscle alone recorded intra-vaginally

Technique to induce fatigue: To apply resistance against contraction of continence muscles and to induce fatigue, the investigators developed a hand-made device in our laboratory; continence muscles resistance device; c-RED . The c-RED consists of a 6 cm x 2 cm noncompliant cylindrical balloon (intra-anal balloon) that is connected to a small compliant balloon (external balloon, about 1.5 x 2 cm) by a 2 mm diameter tube and a stopcock to allow for air to be filled and sealed in the system. To ensure consistent resistance provided by the anal balloon in the study, a commercially available noncompliant valvuloplasty balloon (Z-Med) is chosen to serve as the intra-anal balloon in the c-RED. The system is prefilled with air to determine the amount of air needed for a given internal pressure, or desired resistance of the intra-anal balloon. This is determined using a sphygmomanometer gauge in a sealed system. The intra-anal balloon, while providing resistance, is compressed by the anal contraction (exceeding the internal pressure) due to displacement of its air to the external distensible balloon. The compressibility of the anal balloon allows for the muscle shortening necessary for isotonic exercise. Air displacement into the external balloon results in its expansion allowing to maintain the predetermined intra-anal balloon pressure and serves as an externally visible indicator that an anal contraction has occurred. Using this device, the investigators can choose different level of resistance load on the continence muscles complex (external anal sphincters (EAS) and puborectalis muscle (PRM)).

High-resolution anorectal manometry: Anorectal manometric pressures will be monitored using a high-resolution anorectal manometry catheter (Medical Measurements Systems, Laborie) positioned across the anal canal with the distal end in the rectum. A computerized recording and analysis system stores pressure data from 8 sensor rows (23 pressure sensors total) spaced 1 cm apart along the probe.

High-resolution vaginal manometry: Vaginal pressure recording is a method to record contractile function of the puborectalis muscle. Reliable measurement of the pressure generated by PRM contraction from vaginal cavity has been challenging. However, using a combined technique of Barostat technology and high-resolution Manometry, the investigators have overcome this challenge.

Vaginal Barostat device: This device is commercially available, and its principle of operation is well described previously. Briefly, the investigators applied the capability of the barostat technology to adjust the distending volume in order to achieve the desired pressure against the wall of the hallow organ. The investigators have used this device and method described above.

Methods for detecting PRM contraction: To detect and record the PRM contractile pressure, the investigators used a combined Barostat/high-resolution vaginal manometry technique. Since vaginal canal diameter does not allow necessary contact with the manometric catheter to reliably register contractile activity of the PRM, the investigators used the Barostat technology to provide apposition of the Manometric catheter and vaginal wall and maintaining minimum required contact pressure necessary for sensing and recoding of PRM contraction. Our studies in a group of young female participants (preliminary data) showed that 7-9mmHg pressure was needed to sense the PRM contraction. This set up provides optimal opportunity to record pressure increases induced by PRM short and long-duration contractions.

Method for providing vaginal resistance to PRM contraction: The investigators adapted the c-RED device principle for this purpose. The investigators used vaginal bag (non-stretchable/ non elastic) filled with air providing various intra-bag pressure providing resistance to PRM during Kegel like contractions. To allow compressibility of the bag while maintaining its inner pressure, the investigators connected the bag to a distensible external small balloon similar to the c-RED design described above.

Study subjects: The investigators will study a total of 180 healthy volunteers without past or present history of fecal incontinence in the following age groups: 15 healthy female and 15 healthy males from 6 consecutive decades: 18-30, 31-50, 51-60, 60-70, 70-80, 80 plus years old.

Study Procedure:

To measure the fatigability of continence muscle complex (combined EAS and PRM): subjects will be placed in left lateral position for the duration of the study. Before initiation of the contraction protocol, all subjects will have a digital rectal examination (DRE) and will be asked to perform anal squeezes as instructed during DRE. The investigators ensure that every subject can perform the anal squeezes correctly before initiating the study protocol. The participants will be instructed not to contract their abdomen or buttocks. After applying lubricating gel along the catheter, the high-resolution anorectal manometry catheter will be gently placed inside the anal canal with the distal end in the rectum. This allows for pressure sensors to be arranged along the entire anal canal. After placement of the catheter, a 5-min interval was allotted before the start of the contraction protocol to allow the sphincter tone to return to the basal level. The subjects will be cued to perform Kegel contractions with or without c-RED in place. The sequence will be randomly determined. For contractions with c-RED the anal balloon of the c-RED will be gently placed through the anal canal along the manometric catheter with tip of the anal balloon positioned in the rectum and its distal end visible in the perinium. The anal balloon will then be inflated to achieve the desired resistance pressure of 30, 40 and 50 mmHg pressure (pre-determined pressure randomly selected sequence), as determined with the hand-held pressure gauge. For all contractions participants will be asked to do squeeze anal contraction as hard as possible and hold for 3sec followed by a relaxation time of for 3sec. Participants will be asked to do 40 consecutive squeeze contractions at each pressure level (one set) in a random order. There will be a 5-minutes resting interval between each set. Participants will also perform a long squeeze and hold for 30s at the three above different pressure levels. Participants will do two sustained squeezes separated by 1 minute relaxation period in between.

To measure the fatigability of puborectalis muscle during anal resistive contraction: female subjects will have simultaneous vaginal HRM done during anal squeeze against c-RED. The vaginal barostat bag with HRM catheter attached anteriorly via a sleeve will be gently placed inside the vaginal canal with the distal end of the bag outside the vaginal opening. The vaginal bag will be connected to barostat device to determine the minimum vaginal wall contact pressure to record the PRM contraction as described above.

To measure isolated fatigability of the puborectalis muscle during intra-vaginal resistive contraction: all female subjects will be studied in lithotomy position. The resistance in these experiments will be applied in the vagina rather than anal canal. The manometry probe will be attached to the vaginal barostat bag via a sleeve anteriorly to ensure it is aligned with the vaginal wall when inserted. To provide resistance, the vaginal bag as shown in Figure 8 will be inflated to inner bag pressure of 30, 40 and 50 mmHg. The subjects will be instructed to perform 40 consecutive Kegel type contractions (3sec contraction alternating with 3 sec rest) at the above intra-vaginal pressure levels in random order. There will be a 5-minutes resting interval between each set. Participants will also perform a long squeeze and hold for 30sec at different pressure level. Participants will do two sustained squeezes separated by 1 minute relaxation period in between. Anorectal pressure will be simultaneously recorded by high-resolution Manometry and pressure changes will be correlated to those recorded from the vaginal canal.

Aim 1B: To compare and characterize the differences in fatigue characteristics of the continence muscles induced by isotonic and isometric contractions

Study subjects: same subjects as listed above Aim 1A

Study protocols: These studies will be performed along with studies described in Aim 1A Anal contraction against a non-compressible balloon; Isometric contraction The investigators will use a modified c-RED device for isometric contraction. Our preliminary studies have shown that compressibility of the c-RED is due to the ability of the air to escape from the anal balloon to external balloon, excluding the external balloon from the circuit will prevent air escape which prevents the compressibility of the anal balloon at internal pressures of 500 mmHg. The commercially available balloons used in c-RED is resistant to internal pressures as high as 4 atmosphere (4x760mmHg) far above pressures encountered in these studies. With this arrangement the modified c-RED balloon will provide the anal canal muscles to contract without shortening their length, hence performing isometric contractions. With this approach both isotonic and isometric contractions are done against the same diameter balloon providing comparability of anal canal distension between two types of contractions avoiding potential confounders.

All subjects will be in left lateral position for the duration of the study. After placement of the probe and anorectal manometry catheter, the subjects will be asked to perform 40 consecutive Kegel contractions (3sec contraction alternating with 3sec rest). Participants will also perform long-duration contraction for a period of 30sec. Participants will do three 30sec contractions separated by 1 minute rest period in between.

Anal contraction against compressible balloon; isotonic contraction with c-RED This part will be the same as the studies described in SA1A. Sequence of the two types of contraction studies will be randomized.

Aim 2: Determine the relative/individual contribution of continence muscles (PRM, EAS) motor function enhancement in improving fecal incontinence.

Study subjects: The investigators will study 20 fecal incontinence (FI) patients for each of the eight experimental conditions described below.

Study protocols: Studies will be performed in two steps:

Step 1: This step will serve two purposes; a. to obtain baseline data and b. train the patients on how to perform the contraction protocol at home. This training will be reinforced on a weekly basis through virtual or phone meetings as possible. In this step all participants will undergo baseline studies as described in Aim 1A before starting their at-home contraction protocols. These include baseline resting anal pressure, anal squeeze pressure and vaginal /PRM HPZ pressure (female only). Participants will also undergo fatigue studies as described in Aim 1A. Participants who can perform continence muscles contraction and demonstrate fatigue with the application of the proposed approach at all resistance levels (30, 40 and 50 mmHg) will continue with at-home step 2 protocol.

Step 2: These studies will determine if enhancement of EAS, PRM, or both is required in improving incontinence and in achieving a significant clinical outcome. These studies can be divided in three groups; A. studies using isotonic contractions (protocol 2, 3 & 4) which are aimed to fatigue and are hypothesized to subsequently strengthen: protocol 2. the PRM by 40 Kegel like repetitive short contractions against a progressively increased intra-vaginal resistance (using vaginal c-RED), protocol 3. the EAS by 20 Kegel like repetitive short contractions against a progressively increased intra-anal resistance (using c-RED), protocol 4. combined EAS and PRM by 40 Kegel like repetitive short contractions against a progressively increased intra-anal resistance (using c-RED), B. control studies (protocol 1, 5 &6): protocol 1. will be control for experiment 2; 20 Kegel like repetitive short contractions against a progressively increased intra-vaginal resistance (using vaginal c-RED) and protocol 5 & 6 will serve as controls to experiments 3 & 4 above but without any resistive load, and C. isometric contractions (protocol 7&8): protocol 7. 20 Kegel like repetitive short contractions against the non-compressible balloon described in SA1A and protocol 8. 40 Kegel like short repetitive contractions against the non-compressible balloon described in SA1A. The repetitive short contractions include 3sec contractions followed by 3sec relaxation as described in SA1A. In each of the protocol, participants will perform 3 30sec long contraction as well. Each protocol will be performed twice daily for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without past or present history of fecal incontinence
* Patients age 18 years and older with reduced anal resting and or squeeze pressure, reflecting weakness of the anal sphincters who can perform the study

Exclusion Criteria:

* Any one less than 18 years old
* Neurological disorders like dementia, cerebrovascular diseases
* Muscle diseases like muscular dystrophy, myopathies
* Inflammatory bowel disease or celiac disease
* Neuro-muscular junction disorders/myasthenia gravis, Eaton-Lambert syndrome
* Organ prolapse, large rectocele(>2cm), rectal intussusception
* Hip dysplasia or recent hip surgery and immobile patients.
* Patients with complete normal anal resting and squeeze pressure
* Impaired rectal evacuation (dyssynergy defecation)
* Fecal incontinence completely due to loss of rectal sensation
* Subjects unable to contract their external anal sphincter at all

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
anal pressure | during kegel like exercise
  Maximum squeeze pressure, mean squeeze pressure and anal squeeze contractile integral
anal pressure | after 6 weeks' exercise, during kegel like exercise
  Maximum squeeze pressure, mean squeeze pressure and anal squeeze contractile integral
Vaginal pressure | during kegel like exercise
  Maximum squeeze pressure, mean squeeze pressure and vaginal squeeze contractile integral
Vaginal pressure | after 6 weeks' exercise, during kegel like exercise
  Maximum squeeze pressure, mean squeeze pressure and vaginal squeeze contractile integral
Fecal Incontinence severity | before and after 6 weeks' exercise
  Vaizey Incontinence Score to quantify the severity of fecal incontinence. The Vaizey score is a validated tool and consists of two scoring systems with a five-point scale, which evaluates type and frequency of solid/liquid stool loss, flatus incontinence and impact on quality of life. Vaizey score ranges from 0 to 24, with 0 indicating perfect continent and 24 suggesting complete incontinence.
Quality of life measure | before and after 6 weeks' exercise
  The investigators will use Fecal Incontinence Quality of Life scale (FIQOL).FIQOL is used to evaluate psychometric health-related quality of life parameters in fecal incontinence patients. The score is arranged on four psychosocial scales: lifestyle, coping/behavior, depression/self-perception, and embarrassment, and contains a total of 29 different items. Subscale scores range from 1 to 5 and are the average response to all items on the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mei L, Patel K, Lehal N, Kern MK, Benjamin A, Sanvanson P, Shaker R. Fatigability of the external anal sphincter muscles using a novel strength training resistance exercise device. Am J Physiol Gastrointest Liver Physiol. 2021 Apr 1;320(4):G609-G616. doi: 10.1152/ajpgi.00456.2020. Epub 2021 Feb 17. PMID 33596155
- [Background] Patel K, Mei L, Yu E, Kern M, Lehal N, Edeani F, Sanvanson P, Davidson ERW, Shaker R. Differences in fatigability of muscles involved in fecal continence: Potential clinical ramifications. Physiol Rep. 2021 Dec;9(24):e15144. doi: 10.14814/phy2.15144. PMID 34927399